CLINICAL TRIAL: NCT04140214
Title: A 2x2 Factorial Randomized Open Label Trial to Determine the Clinical and Cost-effectiveness of Hypertonic Saline (HTS) 6% and Carbocisteine for Airway Clearance Versus Usual Care Over 52 Weeks in Bronchiectasis
Brief Title: Randomised Open Label Trial of Hypertonic Saline and Carbocisteine in Bronchiectasis (CLEAR)
Acronym: CLEAR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Belfast Health and Social Care Trust (Other)
Collaborators: Queen's University, Belfast (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 16178SE-AS
Record Dates: First submitted 2019-05-17; First posted 2019-10-25 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-01

CONDITIONS: Bronchiectasis
Keywords: Respiratory; Mucoactive; Exacerbation; Hypertonic Saline; Carbocisteine; Airway Clearance
MeSH Terms: conditions — Bronchiectasis | interventions — Saline Solution, Hypertonic; Carbocysteine

STUDY DESIGN:
Intervention Model Description: A superiority, 2x2 factorial randomised open label trial with a 52-week follow-up period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Standard Care and HTS (Experimental): Standard care and twice-daily nebulised HTS (MucoClear 6%, PARI Pharma). Participants will be instructed to administer a 1 x 4 mL ampoule twice daily for 52 weeks using the eFlow rapid nebuliser and eTrack controller (PARI Pharma).
  Interventions: Drug: Hypertonic saline
- Standard Care and Carbocisteine (Experimental): Standard care and carbocisteine (750 mg three-times-per-day until visit 3, reducing to 750 mg two times per day) over 52 weeks.
  Interventions: Drug: Carbocysteine 750 MG
- Standard Care and Combination of HTS and Carbocisteine (Experimental): Standard care and combination of twice-daily nebulised HTS (MucoClear 6%, PARI Pharma) and carbocisteine. Participants will be instructed to administer a 1 x 4 mL ampoule twice daily for 52 weeks using the eFlow rapid nebuliser eFlow rapid nebuliser and eTrack controller (PARI Pharma). They will also be given carbocisteine (750 mg of three times per day until visit 3, reducing to 750 mg twice per day) over 52 weeks.
  Interventions: Drug: Hypertonic saline; Drug: Carbocysteine 750 MG
- Standard Care Only (No Intervention): Standard care over 52 weeks. Patients in the standard care group will use airway clearance techniques in the management of their BE.

INTERVENTIONS:
Drug: Hypertonic saline — Nebulized hypertonic saline solution (6%)
  Other Names: MucoClear 6%; HTS
  Arms: Standard Care and Combination of HTS and Carbocisteine; Standard Care and HTS
Drug: Carbocysteine 750 MG — Carbocisteine tablet
  Other Names: Mucodyne
  Arms: Standard Care and Carbocisteine; Standard Care and Combination of HTS and Carbocisteine

SUMMARY:
Patients with bronchiectasis (BE) suffer from a persistent cough, daily sputum expectoration, recurrent chest infections, and a poor health-related quality of life. Current guidelines for the management of BE highlight the lack of evidence to recommend mucoactive agents, such as hypertonic saline (HTS) and carbocisteine, to aid sputum-removal as part of standard care. The investigators hypothesise that mucoactive agents (HTS or cabocisteine, or a combination of both) are effective in reducing exacerbations over a 52-week period, compared to usual care.

DETAILED DESCRIPTION:
Mucus hypersecretion is a clinical feature of BE. This mucus-retention aids bacterial infection that can lead to pulmonary exacerbations, which further develops the "viscous cycle" of mucus-retention, infection, inflammation and tissue damage. Mucoactive drugs target this cycle by potentially increasing the ability to expectorate sputum and/or decrease mucus hypersecretion.

The current guidelines indicate that mucoactives in combination with airway clearance may be considered to enhance sputum expectoration in BE, but the evidence to support their use is limited. Furthermore, evidence for the effectiveness of hypertonic saline (HTS) and carbocisteine is insufficient to recommend them within the management of BE. However, EMBARC/BRONCH-UK data show that BE centres do prescribe mucoactives. This is important because adherence to therapies in BE in general is low, decreases as the number of prescribed medications increases, and is also related to poorer patient outcomes, including the number of pulmonary exacerbations and quality of life. Therefore, it is essential that only those drugs that are effective should be prescribed for patients with BE. There are cost considerations associated with mucoactives, and there is a risk of polypharmacy side effects.

Unlike BE, relatively strong evidence exists to favour the use of both HTS and carbocisteine within other respiratory conditions. Therefore, this trial will answer important clinical questions about whether similar benefits can be demonstrated in BE by using a pragmatic design to explore the specific effects of mucoactive agents, and directly support, or refute, more targeted use of these drugs.

Patients will be randomised to one of four treatment groups: (i) standard care and twice daily nebulised HTS (6%), (ii) standard care and carbocisteine, (iii) standard care and combination of twice-daily nebulised HTS and carbocisteine, or (iv) standard care alone.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of BE on high resolution computed tomography(HRCT)/computed tomography (CT) scans
* BE must be the primary respiratory diagnosis
* One or more pulmonary exacerbations in the last year requiring antibiotics*
* Production of daily sputum
* Stable for 14 or more days before the first study visit with no changes to treatment
* Willing to continue any other existing chronic medication throughout the study
* Female subjects must be either surgically sterile, postmenopausal or agree to use effective contraception during the treatment period of the trial *This can include patient reported exacerbations

Exclusion Criteria:

* Age <18 years old
* Patients with cystic fibrosis (CF)
* Patients with COPD as a primary respiratory diagnosis
* Current smokers, female ex-smokers with greater than 20 pack years and male ex-smokers with greater than 25 pack years.
* Forced expiratory volume in one second (FEV1) <30%
* If being treated with long term macrolides, on treatment for less than one month before joining study
* Patients on regular isotonic saline
* Treatment with HTS, carbocisteine or any mucolytics within the past 30 days
* Known contraindication or intolerance to hypertonic saline or carbocisteine
* Hypersensitivity to any of the active ingredients or the excipients of carbocisteine
* Active peptic ulceration
* Any heredity galactose intolerance, the Lapp-Lactase deficiency or glucose-galactose malabsorption
* Patients unable to swallow oral capsules
* Women who are pregnant or lactating
* Participation in other trials of investigational products within 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2018-06-27 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-12-18 (Actual)

PRIMARY OUTCOMES:
Mean Number of Exacerbations | 52 weeks post-randomization
  Patient-reported exacerbations assessed using pre-defined criteria, including intensity and duration of symptoms, via modified Respiratory and Systemic Symptoms questionnaire.

SECONDARY OUTCOMES:
Disease-Specific Health-Related Quality of Life | 52 weeks post-randomization
  Respiratory symptoms domain of quality of life with BE (QoL B) questionnaire.
Time to Next Exacerbation | Over 52 weeks post-randomization
  Exacerbations assessed using pre-defined criteria, including intensity and duration of symptoms, via modified Respiratory and Systemic Symptoms questionnaire.
Number of Days of Antibiotics for Exacerbations | Over 52 weeks post-randomization
  Days of antibiotic use directly related to pulmonary exacerbation; assessed using pre-defined criteria for exacerbations, including intensity and duration of symptoms via modified Respiratory and Systemic Symptoms questionnaire and through interview with participant.
Generic Health-Related Quality of Life (HRQoL) | Assessed at baseline, and 2 weeks, 8 weeks, 26 weeks and 52 weeks post-randomization.
  EQ-ED-5L questionnaire; a validated questionnaire that provides a simple descriptive profile and a single index value for health status.
Health Service Use | 52 weeks post-randomization
  Study-specific health-service use questionnaire to capture service use and details of prescribed medications (including antibiotics).
Quality Adjusted Life Years (QALY) | 52 weeks post-randomization
  Calculated by assessment of generic HRQoL measured using the EQ-5D-5L questionnaire. Responses will be converted to utility scores using the tariff recommended by NICE in their Guide to Technology Appraisal at the time of analysis. Currently this is the Crosswalk Value Set. The area under the curve method will be used to calculate Quality adjusted life years (QALYs).
Measurement of Health Impairment | Assessed at baseline, and 2 weeks, 8 weeks, 26 weeks and 52 weeks post-randomization.
  St. Georges Respiratory Questionnaire; designed to measure health impairment in those with COPD and asthma, and validated for use in the BE population.
  Part 1 : Symptoms component (frequency & severity) with a 1, 3 or 12-month recall (best performance with 3- and 12-month recall); Part 2: Activities that cause or are limited by breathlessness; Impact components (social functioning, psychological disturbances resulting from airways disease) refer to current state as the recall.
  Scores range from 0 to 100, with higher scores indicating more limitations. Scaling of items Part I (Symptoms): several scales; Part II (Activity and Impacts): dichotomous (true/false) except last question (4-point Likert scale)
Patient Preferences for Treatment | Assessed at 2, 8, 26, and 52 weeks post-randomization.
  Measured via the TSQM version II questionnaire to assess four key dimensions of treatment satisfaction: effectiveness; side effects; convenience; and global satisfaction (score 0-100, higher scores indicate better satisfaction).
Number of Adverse Events | Over 52 weeks post-randomization
  Reported by the PI or designee via interview with patients.
Changes in Lung Function | 52 weeks post-randomization
  Spirometry testing to measure lung function parameters, to include FEV1, FVC, FEF25-75 and FEV1% predicted.
IMP Adherence | 52 weeks post-randomization
  Assessed using IMP Accountability Logs
HTS Adherence | 52 weeks post-randomization
  Assessed electronically via tracking of nebulizer use.

CONTACTS AND LOCATIONS:
Overall Officials: J. Stuart Elborn, Principal Investigator — Queen's University, Belfast
Locations (20):
- United Kingdom (20):
  - Stoke Mandeville Hospital, Aylesbury
  - Belfast City Hospital, Belfast Health and Social Care Trust, Belfast
  - Queen Elizabeth Hospital, University Hospital Birmingham NHS Foundation Trust, Birmingham
  - Blackpool Teaching Hospitals NHS Foundation Trust, Blackpool
  - Bradford Teaching Hospitals, Bradford
  - Royal Brompton Hospital, Royal Brompton and Harefield NHS Foundation Trust, Brompton
  - Ninewells Hospital and Medical School, NHS Tayside, Dundee
  - Royal Infirmary Edinburgh, NHS Lothian, Edinburgh
  - Royal Free Hospital, Royal Free London NHS Foundation Trust, Hamstead
  - Princess Alexandra Hospital, The Princess Alexandra Hospital NHS Trust, Harlow
  - Royal Lancaster Infirmary, University Hospitals of Morecambe Bay NHS Foundation Trust, Lancaster
  - Cardiff & Vale University Heath Board, Llandough
  - Altnagelvin Area Hospital, Western Health and Social Care Trust, Londonderry
  - Milton Keynes University Hospital, Milton Keynes
  - Freeman Hospital, The Newcastle Upon Tyne Hospitals NHS Foundation Trust, Newcastle
  - Northumbria NHS Foundation Trust, North Shields
  - Churchill Hospital, Oxford University Hospitals NHS Foundation Trust, Oxford
  - Southampton General Hospital, University Hospital Southampton NHS Foundation Trust, Southampton
  - Royal Gwent Hospital, Aneurin Bevan University Health Board, Wales
  - Sandwell & West Birmingham, West Bromwich

IPD SHARING:
Plan to Share IPD: No
Requests for data sharing will be reviewed on an individual basis by the Chief Investigator (CI) and the Trial Management Group (TMG).